CLINICAL TRIAL: NCT02461199
Title: Prospective Observational Study of Fecal Microbiota Transplantation Used to Eradicate Gut-colonizing Multidrug-resistant Bacteria in Patients With Blood Disorders
Brief Title: Stool Transplantation to Reduce Antibiotic Resistance Transmission
Acronym: START
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Grzegorz W. Basak, Associate Professor, Medical University of Warsaw
Other Study IDs: 02KOHAM
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Blood Disorders
Keywords: Fecal microbiota transplantation; Gut colonization; Multidrug-resistant bacteria; Blood disorders; Drug Resistance, Multiple; Disease Eradication
MeSH Terms: conditions — Hematologic Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples collected before and after the procedure.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fecal microbiota transplantation: Patients with proven gut colonization status with following bacteria: Klebsiella pneumoniae resistant to carbapenems, Pseudomonas aeruginosa resistant to carbapenems, Enterococcus faecalis VRE (vancomycin-resistant enterococcus), Enterococcus faecium VRE, Enterobacter cloacae resistant to carbapenems or other MDR species. Gut colonization proven by conventional microbiological culture and/or molecular methods.
  Interventions: Biological: Fecal microbiota transplantation

INTERVENTIONS:
Biological: Fecal microbiota transplantation — Transplantation of 100 ml of fecal microbiota suspension obtained from healthy unrelated donor in two consecutive days via the nasoduodenal tube
  Other Names: FMT

SUMMARY:
During this prospective observational study, the investigators collect the information about the outcomes of fecal microbiota transplantation in patients with blood disorders, performed to eradicate gut colonization with multidrug-resistant (MDR) bacteria.

Patients with blood disorders are characterized by poor diversity of gut microbiome, affected by repeated chemotherapy and antimicrobial treatments. This makes them vulnerable to colonization by pathogenic bacteria carrying genes responsible for antibiotic resistance. In case of gut mucosa injury and severe immune suppression, these colonizing bacteria may cause severe systemic infections. As the bacteria are secreted with the stool, the colonized patients become an epidemiologic threat to the others.

Fecal microbiota transplantation (FMT) was shown to be very efficient in treatment of relapsed and refractory Clostridium difficile infection and became a standard treatment. In home institution, the investigators use FMT not only in case of Clostridium difficile colitis, but also in case of gut colonization with multidrug-resistant (MDR) bacteria. This is based on assumption that physiological gut flora may outcompete the pathogenic bacteria similarly as in case of Clostridium difficile and lead to loss of colonization. The procedure is performed in all patients colonized, who qualify according to listed inclusion and exclusion criteria .

ELIGIBILITY:
Inclusion Criteria:

* Age >18 y
* Carrier status of MDR bacteria in stool: Klebsiella pneumoniae resistant to carbapenems, Pseudomonas aeruginosa resistant to carbapenems, Enterococcus faecalis VRE, Enterococcus faecium VRE, Enterobacter cloacae KPC+ or other MDR species documented by at least two stool cultures
* Blood neutrophil count > 500/uL on the day of fecal microbiota transplantation

Exclusion Criteria:

* Inability to obtain informed consent and lack of consent
* Blood neutrophil count <500/uL on the day of fecal microbiota transplantation or expected decrease to the mentioned number within 2 consecutive days
* Intensive, myelosuppressive chemotherapy (e.g. DHAP, ICE, ESHAP, HD-Cy, HD-Ara-C, DA, conditioning before allogeneic stem cell transplantation, BEACOPP) planned within 2 consecutive days
* Patients up to 1 month after hematopoietic stem cell transplantation
* Clinical signs of mucositis
* Severe liver failure
* Patients undergoing intensive antimicrobial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with blood disorders treated in the Department of Hematology, Oncology and Internal Diseases, with positive gut colonization status with MDR bacteria, who consent for fecal microbiota transplantation.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Eradication of gut colonizing bacteria as proven by at least two negative stool cultures. | 2 weeks to 6 months after fecal microbiota transplantation

SECONDARY OUTCOMES:
Eradication of gut colonizing bacteria as proven by PCR. | 2 weeks to 6 months after fecal microbiota transplantation
Incidence of infective episodes | from day "0" (day of FMT) to 6 months after fecal microbiota transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Basak, MD, PhD, Principal Investigator — Department of Hematology, Oncology and Internal Diseases, the Medical University of Warsaw; Wieslaw Wiktor-Jedrzejczak, MD, PhD, Study Chair — Department of Hematology, Oncology and Internal Diseases, the Medical University of Warsaw
Locations (1):
- Department of Hematology, Oncology and Internal Diseaes, The Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Bilinski J, Grzesiowski P, Sorensen N, Madry K, Muszynski J, Robak K, Wroblewska M, Dzieciatkowski T, Dulny G, Dwilewicz-Trojaczek J, Wiktor-Jedrzejczak W, Basak GW. Fecal Microbiota Transplantation in Patients With Blood Disorders Inhibits Gut Colonization With Antibiotic-Resistant Bacteria: Results of a Prospective, Single-Center Study. Clin Infect Dis. 2017 Aug 1;65(3):364-370. doi: 10.1093/cid/cix252. PMID 28369341
- [Derived] Bilinski J, Grzesiowski P, Muszynski J, Wroblewska M, Madry K, Robak K, Dzieciatkowski T, Wiktor-Jedrzejczak W, Basak GW. Fecal Microbiota Transplantation Inhibits Multidrug-Resistant Gut Pathogens: Preliminary Report Performed in an Immunocompromised Host. Arch Immunol Ther Exp (Warsz). 2016 Jun;64(3):255-8. doi: 10.1007/s00005-016-0387-9. Epub 2016 Mar 9. PMID 26960790